CLINICAL TRIAL: NCT02928445
Title: A Long-Term Extension Study of the Safety and Tolerability of RVT-101 in Subjects With Dementia With Lewy Bodies (DLB)
Brief Title: Long-Term Extension Study of Intepirdine (RVT-101) in Subjects With Dementia With Lewy Bodies: HEADWAY-DLB Extension
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Intepirdine did not meet its primary efficacy endpoints in the lead-in study RVT-101-2001.
Sponsor: Axovant Sciences Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sio Gene Therapies (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVT-101-2002
Record Dates: First submitted 2016-10-07; First posted 2016-10-10 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-02

CONDITIONS: Dementia With Lewy Bodies
Keywords: Dementia with Lewy bodies; dementia; RVT-101; intepirdine; Lewy bodies
MeSH Terms: conditions — Lewy Body Disease; Dementia | interventions — 3-benzenesulfonyl-8-piperazin-1-ylquinoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RVT-101 35 mg (Experimental): RVT-101 35 mg once daily
  Interventions: Drug: RVT-101 35 mg
- RVT-101 70 mg (Experimental): RVT-101 70 mg once daily
  Interventions: Drug: RVT-101 70 mg

INTERVENTIONS:
Drug: RVT-101 35 mg — once daily, oral, 35-mg tablets
  Arms: RVT-101 35 mg
Drug: RVT-101 70 mg — once daily, oral, 35-mg tablets
  Arms: RVT-101 70 mg

SUMMARY:
This 6-month extension study will provide further information regarding the long-term safety and tolerability of intepirdine (RVT-101) in subjects with Dementia with Lewy bodies (DLB) who have participated in the double-blind, placebo-controlled, lead-in study RVT-101-2001.

DETAILED DESCRIPTION:
This 6-month, double-blind,extension study will provide further information regarding the long-term safety and tolerability of intepirdine (RVT-101) in subjects with DLB who have participated in the double-blind, placebo-controlled, lead-in study RVT-101-2001. The study duration for subjects in study centers in the USA will be 12 months.

Subjects who were randomized to the RVT-101 35-mg and RVT-101 70-mg treatment groups in lead-in study RVT-101-2001 will remain in the same treatment groups for this study; subjects who were randomized to the placebo treatment group in the lead-in study will be assigned to the RVT-101 70-mg treatment group in this study.

Various background therapies, including acetylcholinesterase inhibitors and memantine, will be allowed.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the lead-in study RVT-101-2001.

Exclusion Criteria:

* Any clinically relevant concomitant disease, which, in the opinion of the Investigator, makes the subject unsuitable for inclusion in the study.

Ages: 50 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and changes in physical examinations, vital sign measurements, electrocardiograms (ECGs), and clinical laboratory assessments | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ilise Lombardo, MD, Study Director — Axovant Sciences Inc., Senior Vice President, Clinical Research
Locations (56):
- United States (27):
  - US138, Phoenix, Arizona
  - US108, Phoenix, Arizona
  - US139, Sun City, Arizona
  - US125, Tucson, Arizona
  - US119, Orange, California
  - US134, Oxnard, California
  - US133, Rancho Mirage, California
  - US140, Sacramento, California
  - US141, Englewood, Colorado
  - US123, Washington D.C., District of Columbia
  - US104, Boca Raton, Florida
  - US111, Jacksonville, Florida
  - US122, Orlando, Florida
  - US137, Palm Beach Gardens, Florida
  - US126, Tampa, Florida
  - US136, Atlanta, Georgia
  - US118, Indianapolis, Indiana
  - US105, Lexington, Kentucky
  - US130, Quincy, Massachusetts
  - US102, Rochester, Minnesota
  - US109, New York, New York
  - US100, Chapel Hill, North Carolina
  - US110, Cleveland, Ohio
  - US106, Columbus, Ohio
  - US131, Portland, Oregon
  - US120, Willow Grove, Pennsylvania
  - US101, Charlottesville, Virginia
- CA200, Toronto, Ontario, Canada
- France (8):
  - FR952, Toulouse, Haute-Garonne
  - FR957, Lille, Nord
  - FR951, Villeurbanne, Rhone
  - FR959, Paris
  - FR960, Paris
  - FR953, Saint-Herblain
  - FR950, Strasbourg
  - FR955, Vandœuvre-lès-Nancy
- Italy (6):
  - IT304, Tricase, Lecce
  - IT300, Genoa, Liguria
  - IT302, Brescia, Lombardy
  - IT306, Brescia
  - IT301, Milan
  - IT305, Venice
- Netherlands (2):
  - NE402, Amsterdam, North Holland
  - NE401, 's-Hertogenbosch
- Spain (2):
  - SP600, Barcelona
  - SP605, Barcelona
- United Kingdom (10):
  - UK801, Cambridge, Cambridgeshire
  - UK808, Epping, Essex
  - UK804, Southampton, Hampshire
  - UK807, Bristol
  - UK806, Dundee
  - UK805, Isleworth
  - UK800, London
  - UK809, London
  - UK802, Manchester
  - UK803, Newcastle upon Tyne